CLINICAL TRIAL: NCT06051578
Title: Abdominal Wall Tension in Patients Undergoing Ventral Hernia Repair Without Component Separation
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Benjamin T. Miller, Principal Investigator, The Cleveland Clinic
Other Study IDs: 23-857
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hernia, Ventral; Hernia, Abdominal; Hernia Abdominal Wall
MeSH Terms: conditions — Hernia, Ventral; Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Abdominal wall tension measurement — All patients will have the tension of their abdominal wall measured during surgery using a tension scale or "tensiometer."

SUMMARY:
The purpose of this study is to use a scale to learn more about the tension of the abdominal wall in hernia repairs without component separation.

1. What is the abdominal wall tension for hernias repaired without a component separation?
2. What patient factors contribute to greater abdominal wall tension?
3. Is there an association between abdominal wall tension before primary closure or bridging repair and patient outcomes?

Participants will be asked to allow their surgeon to use a tension scale to measure the tension of the abdominal wall during surgery.

DETAILED DESCRIPTION:
This is a prospective cohort study. Patients who undergo hernia repair without component separation will have their abdominal wall tension measured using a tension scale. The scale is an investigational (experimental) device that works by attaching to surgical clamps during surgery to measure the tension on the abdominal wall. The study operations will be performed at Cleveland Clinic by six hernia surgeons with advanced abdominal wall reconstruction training.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are planned to undergo ventral hernia repair without component separation
2. Midline hernia

Exclusion Criteria:

1. Mesh excision for reasons other than mesh infection
2. Prior component separation
3. Isolated flank hernia
4. Patients under the age of 18 years
5. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 50 patients who have been evaluated by a surgeon and will undergo a hernia repair without component separation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal wall tension in patients hernia repair without component separation | 2 year
  The abdominal wall tension prior to closure will be measured

SECONDARY OUTCOMES:
Patient factors that contribute to greater abdominal wall tension | 2 year
  Patient demographics, comorbidities, operative history, operative details, hernia size and width and abdominal wall tension will be collected and analyzed to determine what factors contribute to abdominal wall tension.
Association between abdominal wall tension and patient outcomes | 2 year
  Abdominal wall tension will be determined and patient outcomes will be analyzed including complications, wound morbidity, recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Miller, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No